CLINICAL TRIAL: NCT00004571
Title: Structural and Functional Imaging of Neuropsychiatric Patients and Normal Volunteers With 3.0 Tesla MRI and Magnetoencephalography (MEG)
Brief Title: Magnetic Resonance Imaging (MRI) of Neuropsychiatric Patients and Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000085; 00-M-0085
Record Dates: First submitted 2000-02-15; First posted 2000-02-16 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-09-09

CONDITIONS: Schizophrenia; Normal Physiology
Keywords: fMRI; MEG; Cognition; Magnetic Resonance Imaging; Schizophrenia; Natural History
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy volunteers: Healthy subjects from the community
- Schizophrenia: Patients with schizophrenia and psychosis
- Williams Syndrome: Individuals with copy number variation in the Williams Syndrome Region

SUMMARY:
The purpose of this study is to use brain imaging technology to compare differences in brain structure, chemistry, and functioning in individuals with brain and mental disorders compared to healthy volunteers.

Schizophrenia is a brain disorder that results from subtle changes and abnormalities in neurons. These deficits likely occur in localized regions of the brain and may result in widespread, devastating consequences. The neuronal abnormalities are inherited through a complex combination of genetic and environmental factors. Brain imaging technologies can be used to better characterize brain changes in individuals with schizophrenia. This study will use magnetic resonance imaging (MRI) scans to identify predictable, quantifiable abnormalities in neurophysiology, neurochemistry and neuroanatomy that characterize schizophrenia and other neurological and neuropsychiatric disorders.

DETAILED DESCRIPTION:
This protocol is meant to provide a matrix for multiple, simultaneous brain imaging investigations using magnetic resonance imaging (MRI) at 3.0 Tesla (3T). We intend to study regional brain structure, physiology, and biochemistry in living human subjects, both healthy and ill. Based on multiple clinical, neuropathological, and functional neuroimaging studies, it is clear that schizophrenia is a brain disorder arising from subtle neuronal deficits (for lack of more specific terminology). These deficits likely arise in a few key regions such as dorsolateral prefrontal cortex and hippocampal formation, that result in widespread, multifaceted, and devastating clinical consequences. These neuronal deficits are clearly heritable, although in a complex fashion from multiple genes interacting in an epistatic fashion with each other and the environment. We hypothesize that these neuronal deficits, clearly resulting in quantifiable behavioral abnormalities in schizophrenic patients, will produce predictable, quantifiable aberrations in neurophysiology that we can "map" using magnetic resonance imaging. In spite of numerous functional imaging findings, clinical applications remain scarce and pathognomonic findings absent. Therefore, we do not anticipate that an approach based solely on any one modality is likely to significantly advance our knowledge base. Instead, we propose to create brain imaging datasets for individual human subjects predicated on 1) the appraisal of brain function from multiple domains simultaneously; 2) the characterization of brain function via summation and intercorrelation of these data; and 3) the digestion of these data based on the parsing of complex clinical phenomenology into quantifiable neurophysiological parameters. Thus, in addition to the identification of those parameters that best characterize and identify manifest schizophrenia (i.e., state variables), we hypothesize that some of these fundamental characteristics will be heritable. These fundamental characteristics, so-called endo- or intermediate phenotypes, represent powerful tools to find susceptibility genes and have already generated a number of linkage findings.

ELIGIBILITY:
* INCLUSION CRITERIA:

CONTROLS:

No psychiatric or severe chronic medical illness at the time of the study, and by history. This includes the absence of substance abuse histories, learning disabilities and all DSM IV disorders. The investigators will evaluate medical histories and medical conditions that are judged not to interfere with the study may be allowed.

No use of psychotropic substances in the last 3 months.

There is no upper age limit. The lower age limit is 18 years.

Controls will all have the capacity to consent.

PATIENTS:

Schizophrenia, any subtype or schizo-affective disorder according to DSM IV .

Bipolar Disorder with Psychotic Features according to DSM IV.

Menstrually-Related Mood Disorder.

Mild to Moderate Parkinson's Disease (Hoehn and Yahr Stage 1-3).

Williams Syndrome (partial or full) with IQ in the normal range.

Patients with Multiple Sclerosis.

EXCLUSION CRITERIA:

CONTROLS AND PATIENTS:

Impaired hearing.

Pregnancy.

Head trauma with loss of consciousness in the last year, or any evidence of functional impairment due to and persisting after head trauma.

Patients or healthy volunteers with a known risk from exposure to high magnetic fields (e.g. patients with pace makers) and those who have metallic implants (e.g. braces) in the head region (likely to create artifact on the MRI scans) will be excluded from participating in the fMRI studies.

History of any (excepting nicotine-related) DSM5-defined moderate to severe substance use disorder (or DSM-IV-defined substance dependence).

Cumulative lifetime history of any (excepting nicotine-related) DSM5-defined mild substance use disorder (or any DSM-IV-defined substance abuse), either in excess of 5 years total or not in remission for at least 6 months.

NIMH employees and staff and their immediate family members will be excluded from the study per NIMH policy.

Non-NIMH NIH employees and staff may participate and will be given the NIH Frequently Asked Questions (FAQs) for NIH Staff Who are Considering Participation in NIH Research.

PATIENTS:

Coexistence of another major mental illness at the time of the study. If the patients experienced other mental illnesses in the past (e.g. a learning disability or major depression), then this should be judged to be fully recovered.

Major concurrent medical illness likely to interfere with the acquisition of the task.

Concomitant medications which could interfere with performance on the task.

Involuntary movements that interfere with positioning in the MRI scanner).

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with schizophrenia and healthy subjects from the community.
Sampling Method: Non-Probability Sample
Enrollment: 3273 (Actual)
Dates: Start 2000-02-17 (Actual)

PRIMARY OUTCOMES:
regional MRSI measures | spectroscopy
  GABA and glutamate measurements in schizophrenia and healthy controls.
magnetic field potentials | MEG
  Group differences in MEG signal for patients with schizophrenia and healthy subjects.
fMRI BOLD responses | MRI study completion
  Group differences between patients with schizophrenia and healthy subjects, also genotyping used to characterize subjects as well.
DTI anisotropy measures | DTI
  Compare fractional anisotropy and other measures of white matter connectivity for schizophrenic patients and controls.
brain volumetric measures | VBM
  VBM and cortical parcellation are used in schizophrenia and healthy controls.

SECONDARY OUTCOMES:
neuropsychological task performance data | NPT

CONTACTS AND LOCATIONS:
Overall Officials: Karen F Berman, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Ianni AM, Eisenberg DP, Boorman ED, Constantino SM, Hegarty CE, Gregory MD, Masdeu JC, Kohn PD, Behrens TE, Berman KF. PET-measured human dopamine synthesis capacity and receptor availability predict trading rewards and time-costs during foraging. Nat Commun. 2023 Sep 30;14(1):6122. doi: 10.1038/s41467-023-41897-0. PMID 37777515
- [Derived] Kippenhan JS, Gregory MD, Nash T, Kohn P, Mervis CB, Eisenberg DP, Garvey MH, Roe K, Morris CA, Kolachana B, Pani AM, Sorcher L, Berman KF. Dorsal visual stream and LIMK1: hemideletion, haplotype, and enduring effects in children with Williams syndrome. J Neurodev Disord. 2023 Aug 26;15(1):29. doi: 10.1186/s11689-023-09493-x. PMID 37633900
- [Derived] Rubinstein DY, Eisenberg DP, Carver FW, Holroyd T, Apud JA, Coppola R, Berman KF. Spatiotemporal Alterations in Working Memory-Related Beta Band Neuromagnetic Activity of Patients With Schizophrenia On and Off Antipsychotic Medication: Investigation With MEG. Schizophr Bull. 2023 May 3;49(3):669-678. doi: 10.1093/schbul/sbac178. PMID 36772948
- [Derived] Marenco S, Meyer C, van der Veen JW, Zhang Y, Kelly R, Shen J, Weinberger DR, Dickinson D, Berman KF. Role of gamma-amino-butyric acid in the dorsal anterior cingulate in age-associated changes in cognition. Neuropsychopharmacology. 2018 Oct;43(11):2285-2291. doi: 10.1038/s41386-018-0134-5. Epub 2018 Jul 3. PMID 30050047
- [Derived] Jabbi M, Cropp B, Nash T, Kohn P, Kippenhan JS, Masdeu JC, Mattay R, Kolachana B, Berman KF. BDNF Val66Met polymorphism tunes frontolimbic circuitry during affective contextual learning. Neuroimage. 2017 Nov 15;162:373-383. doi: 10.1016/j.neuroimage.2017.08.080. Epub 2017 Sep 1. PMID 28867340
- [Derived] Wei SM, Baller EB, Kohn PD, Kippenhan JS, Kolachana B, Soldin SJ, Rubinow DR, Schmidt PJ, Berman KF. Brain-derived neurotrophic factor Val66Met genotype and ovarian steroids interactively modulate working memory-related hippocampal function in women: a multimodal neuroimaging study. Mol Psychiatry. 2018 Apr;23(4):1066-1075. doi: 10.1038/mp.2017.72. Epub 2017 Apr 18. PMID 28416813
- [Derived] Jabbi M, Chen Q, Turner N, Kohn P, White M, Kippenhan JS, Dickinson D, Kolachana B, Mattay V, Weinberger DR, Berman KF. Variation in the Williams syndrome GTF2I gene and anxiety proneness interactively affect prefrontal cortical response to aversive stimuli. Transl Psychiatry. 2015 Aug 18;5(8):e622. doi: 10.1038/tp.2015.98. PMID 26285132
- [Derived] Jabbi M, Kohn PD, Nash T, Ianni A, Coutlee C, Holroyd T, Carver FW, Chen Q, Cropp B, Kippenhan JS, Robinson SE, Coppola R, Berman KF. Convergent BOLD and Beta-Band Activity in Superior Temporal Sulcus and Frontolimbic Circuitry Underpins Human Emotion Cognition. Cereb Cortex. 2015 Jul;25(7):1878-88. doi: 10.1093/cercor/bht427. Epub 2014 Jan 23. PMID 24464944
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2000-M-0085.html